CLINICAL TRIAL: NCT04498442
Title: A Study on Prevalence, Protection and Recovery From COVID-19 in Seasoned Yoga Practitioners in Comparison to Age and Gender Matched Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, PI, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P000433
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Stress; Anxiety Depression
Keywords: covid-19; yoga; stress; anxiety; depression; well being; resilience; breathing exercises
MeSH Terms: conditions — COVID-19; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: In this prospective randomized control trial, the effects of yoga practices are being compared between seasoned yoga practitioners with two controls who are age and gender matched and living in the same neighborhood.
  One control group acts as active control who receives active intervention in the form of yoga activities during the study duration. The study provides its active control group an opportunity to learn and practice Simha-Kriya which involves deep breathing exercises and meditation. In contrast, the other control group acts as a placebo control and performs either reading activities or remains idle for 15 minutes throughout the study period.
  The participants will be requested to complete a set of surveys as a part of the research activity. These surveys include validated scales on stress, resilience and well-being; and objective questions on COVID-19 infection and medical history.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Practitioners (No Intervention): Yoga practitioners arm is the observational arm of the study, wherein participants who follow Isha school of yoga and have completed either of the three courses : Inner Engineering Online (IEO), Inner Engineering Completion (Shambhavi Mahamudra kriya) or Shakthi Chalana Kriya can be included in this group. The participant are advised to continue with their routine yoga practice with no change in the duration of practice or frequency of their practices. Participants of this group have expertise in yoga practice and have been practicing yoga for more than 6 weeks before study enrollment.
- Control Yoga (Active Comparator): Control Yoga is the active comparator arm of the study. Participants who are randomly allocated to this group, practice "Simha Kriya", a deep breathing exercise taught by the Isha School of yoga.
  Interventions: Behavioral: Simha Kriya
- Control Idle (Placebo Comparator): Control Idle is the active comparator arm of the study. Participants who are randomly allocated to this group, are advised to either read a book for 15 minutes each day or sit idle for 15 minutes. This is the true control group for the study
  Interventions: Behavioral: Reading a Book

INTERVENTIONS:
Behavioral: Simha Kriya — Simha-Kriya involves deep breathing exercises and meditation. It is the practice of extending the breath, expanding our lung capacity and mental concentration and energizing the body. Simha Kriya, when practiced intentionally will unite the mental, physical, and spiritual body through the breath. For the purpose of this study we advocate practice of Simha Kriya at least once a day.
  Arms: Control Yoga
Behavioral: Reading a Book — Reading a book regularly promotes knowledge enhancement, reduces stress and enhances memory among other benefits. Reading a book is often inculcated into mindfulness research due to it's impact on the personality and attitude. The simple act of reading a book can have a significant impact on their attitudes and can help them cope better with stress. For the purpose of this study, we advocate reading any book/ journal of participants choice routinely for 15 minutes each day. Reading a book could potentially be substituted with sitting idle for 15 minutes if participants wishes to.
  Arms: Control Idle

SUMMARY:
The study is a randomized controlled trail with an observational arm and aims at collecting information on the prevalence of COVID 19 infection in seasoned yoga practitioners by comparing it with the prevalence of COVID-19 infection prevalence rates among age and gender matched control participants who do not practice yoga.

The study hypothesizes that yoga practice promotes protection and enhances recovery from the COVID-19 infection. To prove the hypothesis, the study investigators are collecting and comparing responses from seasoned yoga practitioners to age and gender matched controls participants (who do not practice yoga routinely) regarding their recovery from the COVID 19 infection. Based on validated questionnaires on perceived stress, anxiety, depression, well-being, mindfulness, joy disposition, and resilience in participants over the study duration, the investigators also collect information on participant's mental and emotional predispositions.

DETAILED DESCRIPTION:
Background:

Globally, COVID-19 has resulted in more than 3 million confirmed cases with a continuing rise in numbers. Following the first case detection in the United States on January 20, 2020, there has been a steady rise in the reported cases resulting in all 50 states being affected by the disease. As of April 28, 2020, two million deaths globally have been attributed to this disease. This is an ongoing pandemic, and our understanding of it is continually evolving.

Measures such as social distancing and working remotely have been enforced worldwide to curb disease transmission. This has led to an increased number of people staying indoors and living a more sedentary lifestyle. Many clinicians and people in the community have raised concerns about maintaining good mental and emotional health along with physical health.

Amidst concerns for maintenance of holistic health, yoga in its forms of guided breathing, meditation, and mindfulnessare interventions people are practicing rigorously in the current times of uncertainty. These interventions require no external infrastructure, promote a sense of calm and well-being, improve sleep quality, and reduce stress and anxiety.

Need for the study:

The study aims at collecting information on the prevalence of COVID 19 infection in seasoned yoga practitioners and comparing it with the prevalence of COVID-19 infection prevalence rates among age and gender matched control participants.

The study hypothesizes that yoga practice promotes protection and enhances recovery from the COVID-19 infection. To prove the hypothesis, the study investigators intend to collect and compare responses from seasoned yoga practitioners and age and gender matched controls regarding their recovery from the COVID 19 infection. Based on validated questionnaires on perceived stress, anxiety, depression, well-being, mindfulness, joy disposition, and resilience in participants over the study duration, the study investigators also intend to collect information on participant's mental and emotional predispositions.

Through this Randomized Controlled Trial, the following specific aims are to be accomplished:

Specific Aim 1: To compare prevalence rates of diagnosed COVID-19 infection between the seasoned yoga practitioners and age and gender matched controls at baseline and at 6 and 12 weeks.

Specific Aim 2: To Compare Protection and Recovery from COVID 19 infection between seasoned yoga practitioners and controls as demonstrated by:

1. Self-reported duration of fever and respiratory symptoms in COVID-19 positive participants
2. Self-reported readiness to return to work (or a feeling of being physically and mentally fit) This is the key secondary outcome of the study.

Specific aim 3: To quantitatively assess the effects of yoga practices between seasoned practitioners and the control groups on measures such as perceived stress, resilience, and overall wellbeing by use of validated scales.

We also aim to do exploratory analysis by comparing the different yoga practices and their duration between the 3 study groups to establish a dose-response curve if possible.

Note: The term "yoga" used throughout this document is defined as mindfulness practices which involve deep breathing exercises and meditation, and excludes strenuous physical exercise.

ELIGIBILITY:
Inclusion Criteria:

For Seasoned Yoga practitioners:

* Participants must be a follower of Isha school of yoga
* Must have completed Inner Engineering Online course/ practice Shambhavi Mahamudra Kriya/ Shakthi Chalana Kriya
* Interest in participating in the study

For Controls:

* Participants has little to no experience with Isha school of yoga
* Should have practiced yoga routinely for < 1 Month (if previously experienced in yoga)
* Interest in participating in the study
* Age ( +/- 3 years) matched with the seasoned practitioner
* Gender matched with seasoned practitioner

Exclusion Criteria:

For both groups:

* Participants < 18 years of age
* Participant > 80 years of age
* Participants must be able to read and understand English.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8519 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Levels | Baseline, 6 weeks and 12 weeks.
  The study aims to evaluate changes in perceived levels of stress in survey participants and the effect yoga or reading a book has over them. We use a validated scale for this purpose named, Perceived Stress Scale. The scale measures the degree to which situations in participant's life are appraised as stressful. This is the primary outcome for our study. We assess for change in perceived stress levels by analyzing the PSS score for each participant and comparing it to pre & post intervention results.

SECONDARY OUTCOMES:
Changes in Resilience Levels | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in resilience levels in survey participants and the effect yoga or reading a book has over them. We use a validated scale for this purpose named, Brief Resilience Scale. The scale identifies the individual's ability to bounce back or recover from a stress. This is the key secondary outcome for our study. We assess for change in resilience levels by analyzing the 6-item BRS, which computes a score for each participant by dividing total score obtained/number of questions responded; (range 6-30) and comparing it to pre & post intervention results.
Changes in Covid-19 Prevalence | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in Covid-19 prevalence in survey participants and the effect yoga or reading a book has over them. Based on the reported number of cases in the participant cohort we compute Period Prevalence for 3 specified time points. We assess for change in reported prevalence and stratify the results to match with region-wise prevalence.
Changes in self-reported duration of fever and respiratory symptoms in COVID-19 positive participants | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in self-reported duration of fever and respiratory symptoms in Covid-19 positive survey participants and the effect yoga or reading a book has over them. Based on the reported number of positive cases in the participant cohort we compare the frequency of duration between the two cohorts i.e. yoga practitioners and control; followed by a comparison between the two control groups viz: yoga group vs idle group.
Changes in self-reported readiness to return to work in COVID-19 positive participants | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in self-reported readiness to return to work in Covid-19 positive survey participants and the effect yoga or reading a book has over them. Based on the reported number of positive cases in the participant cohort we compare the frequency of readiness between the two cohorts i.e. yoga practitioners and control; followed by a comparison between the two control groups viz: yoga group vs idle group.

OTHER OUTCOMES:
Changes in Mindfulness | Baseline, 6 weeks and 12 weeks
  We assessed for change in Mindfulness levels in all participants by using a short form of the validated scale for this purpose namely, Mindfulness Attention Awareness Scale (MAAS). The scale measures the individuals' ability for receptive awareness and attention to present. We compute the MAAS scores for each participant which is a mean score for 5 item questionnaires and compare the pre & post intervention results to look for change.
Changes in Dispositional Positive Emotions Scale (DPES- Joy subscale) | Baseline, 6 weeks and 12 weeks
  We assess for change in the individuals' ability to feel joy and look for it in the mundane by using a validated scale for this purpose namely, Dispositional Positive Emotions Scale (DPES) particularly the Joy subscale. The Sub-scale measures the individuals' dispositional ability to feel joy in life. We compute the DPES-JOY subscale scores for each participant which is a mean score for 6 item questionnaires and compare the pre & post intervention results to look for change.
Changes in 4 Item-Patient Health Questionnaire measuring Anxiety and Depression (PHQ-4) levels | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in anxiety and depression levels in survey participants and the effect yoga or reading a book has over them. We use a validated scale for this purpose named, 4 Item-Patient Health Questionnaire measuring Anxiety and Depression (PHQ-4) Scale. The 4 question scale screens for anxiety and depression in participants by computing sum for the responses (scores range: 0-12) and comparing it to pre & post intervention results.
Changes in well being levels | Baseline, 6 weeks and 12 weeks
  The study aims to evaluate changes in wellbeing levels in survey participants and the effect yoga or reading a book has over them. We use a validated scale for this purpose named, Warwick- Edinburgh Wellbeing Scale (WEMWBS). The scale identifies the individual's aspects of mental health such as: positive affect, satisfying interpersonal relationship and positive functioning. We assess for change in 14 item well-being levels by analyzing the total WEMWBS score for each participant and comparing it to pre & post intervention results.
Changes in Post Traumatic Growth Inventory (PTGI) scores | Baseline, 6 weeks and 12 weeks
  The purpose of the growth inventory is to capture the positive outcomes reported by a person who have experienced a traumatic event. This scale collects information from only those participants who identify as being hospitalized during the COVID-19 pandemic and look for their coping ability to the aftermath of the trauma. This 21 item scale is rated on a 6-point Likert response scale. Response from each of the 6 question is then summed to create a total PTGI score.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Upadhyay P, Narayanan S, Khera T, Kelly L, Mathur PA, Shanker A, Novack L, Perez-Robles R, Hoffman KA, Sadhasivam SK, Subramaniam B. Perceived Stress, Resilience, and Wellbeing in Seasoned Isha Yoga Practitioners Compared to Matched Controls During the COVID-19 Pandemic. Front Public Health. 2022 Jul 29;10:813664. doi: 10.3389/fpubh.2022.813664. eCollection 2022. PMID 35968476